CLINICAL TRIAL: NCT02513836
Title: Development of an Innovative Opioid Safety Program in Pain Clinics (Op-Safe): A Multi-Centre Project
Brief Title: Opioid Safety Program in Pain Clinics (Op-Safe):
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dr. Frances Chung, Anesthesiologist, University Health Network, Toronto
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Version: August 17, 2016
Record Dates: First submitted 2015-05-27; First posted 2015-08-03 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Sleep Disordered Breathing
Keywords: opioids
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-education intervention (Experimental): All study participants will be tested with a questionnaire (POEM; Patient Opioids Education Measurement) on their opioid knowledge during 1st visit at the pain clinic.
  Interventions: Other: Pre-education intervention
- Post-education intervention (Other): All study participants will be educated on opioids via an education sheet, pamphlet and video from the Institute for Safe Medication Practices (ISMP) Canada. They will repeat the questionnaire (POEM) after this education on opioid knowledge on the same day.
  Interventions: Other: Post-education intervention

INTERVENTIONS:
Other: Pre-education intervention — All study participants will be tested with a questionnaire (POEM; Patient Opioids Education Measurement) on their opioid knowledge during 1st visit at the pain clinic.
  Arms: Pre-education intervention
Other: Post-education intervention — All study participants will be educated on opioids via an education sheet, pamphlet and video from the Institute for Safe Medication Practices (ISMP) Canada. The questionnaire (POEM) will be tested again after this education on opioid knowledge on the same day.
  Arms: Post-education intervention

SUMMARY:
In this vital study, the investigators will develop an innovative Opioid Safety (Op-Safe) Program for use in pain clinics. The Op-Safe Program consists of two key components: Educating patients with an informative brochure and video developed by the Institute for Safe Medication Practices (ISMP) Canada, and a screening algorithm to identify unrecognized sleep apnea in patients taking opioids for chronic non-cancer pain.

DETAILED DESCRIPTION:
This 2-year prospective multi-centre cohort study will be conducted at chronic pain clinics at Women's College Hospital (WCH), Toronto Western Hospital (TWH), Toronto Rehab Institute (TRI), Mount Sinai Hospital (MSH) in Toronto, and St. Joseph's Hospital (SJH) in London, Ont.

The primary aim is to develop and evaluate an Obstructive Sleep Apnea (OSA) screening algorithm against the results of polysomnography.The research assistants will approach all patients visiting chronic pain clinics for eligibility. For recruited patients, a written informed consent will be obtained. All recruited patients will undergo polysomnography at the Toronto Rehab Institute Sleep Lab or Toronto Sleep and Pulmonary Centre. An overnight oximetry by an oximeter will be collected. The sleep physician will review the polysomnography results.

All recruited patients will also complete the STOP-Bang questionnaire and Epworth Sleepiness Scale (ESS). The thyromental distance, Mallampati classification, Friedman staging,neck circumference and oxygen saturation will be measured. Demographic data, co-morbidities, medications and an overnight oximetry will be collected.

Patients will be assessed on their opioid-related knowledge via the Patient Opioid Education Measure (POEM) at the first visit. They will be educated on knowledge of opioids via education sheet, pamphlet and video from ISMP-Canada, and then repeat Patient Opioid Education Measure (POEM) 6- 8 months later during pain clinic follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥18 years old) with cognitive capability to comprehend the educational intervention who are taking opioid medication for >3 months for non-cancer pain.

Exclusion Criteria:

1. Patients with chronic pain secondary to a neoplasm or metastasis as goals of care are different in this patient population.
2. Patients requiring urgent sleep physician referral (within four weeks) due to serious medical conditions or safety critical-occupations according to the 2011 Canadian Thoracic Society (CTS) guidelines[60] e.g. unstable ischemic heart disease, recent cerebrovascular disease, congestive heart failure, refractory systemic hypertension, pulmonary hypertension, hypercapnic respiratory failure or pregnancy.
3. Conditions potentially interfering with comprehension and delivery of informed consent or the educational intervention, such as neurological or psychiatric disorders.
4. Patients with a prior diagnosis of sleep-related breathing disorder within the last 3 years with treatment. Patients who may have had sleep studies 3 or more years earlier may be included, if they have been lost to follow-up by a sleep physician, are not on treatment or are non-compliant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Predictive performance of screening algorithm for sleep disordered breathing | 30 days
  Predictive performance (sensitivity, specificity, positive predictive value, negative predictive value, and the area under receiver operating characteristic [ROC] curve) of screening algorithm for sleep disordered breathing. A paired t-test will be used to evaluate the changes in opioid related knowledge.

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - London Health Sciences Centre, London, Ontario
  - Toronto Rehab Institute (TRI), Toronto, Ontario
  - Women's College hospital, Toronto, Ontario
  - Toronto Western Hopsital, Pain Clinic, Dept. of Anesthesia, Toronto, Ontario
  - Mount Sinai Hospital, Wasser pain management clinic, Toronto, Ontario

REFERENCES:
- [Derived] Selvanathan J, Waseem R, Peng P, Wong J, Ryan CM, Chung F. Simple screening model for identifying the risk of sleep apnea in patients on opioids for chronic pain. Reg Anesth Pain Med. 2021 Oct;46(10):886-891. doi: 10.1136/rapm-2020-102388. Epub 2021 Aug 9. PMID 34373347
- [Derived] Wasef S, Mir S, Ryan C, Waseem R, Bellingham G, Kashgari A, Wong J, Chung F. Treatment for patients with sleep apnea on opioids for chronic pain: results of the OpSafe trial. J Clin Sleep Med. 2021 Apr 1;17(4):819-824. doi: 10.5664/jcsm.9064. PMID 33382032
- [Derived] Chung F, Wong J, Bellingham G, Lebovic G, Singh M, Waseem R, Peng P, George CFP, Furlan A, Bhatia A, Clarke H, Juurlink DN, Mamdani MM, Horner R, Orser BA, Ryan CM; Op-Safe Investigators. Predictive factors for sleep apnoea in patients on opioids for chronic pain. BMJ Open Respir Res. 2019 Dec 23;6(1):e000523. doi: 10.1136/bmjresp-2019-000523. eCollection 2019. PMID 31908788